CLINICAL TRIAL: NCT06885567
Title: A Multicenter, Randomized, Double-blind, Parallel Design, Placebo-controlled, Phase 2 Clinical Trial and Open-Label Extension Study to Evaluate the Safety and Efficacy for BEY2153 in Patients with Early Alzheimer's Disease
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of BEY2153 in Patients with Early Alzheimer's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BeyondBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BEY-2022-01
Record Dates: First submitted 2025-03-10; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease; Alzheimer' Disease
MeSH Terms: conditions — Alzheimer Disease; Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- BEY2153 dose 1 (Experimental): Participants administer 26 weeks
  Interventions: Drug: BEY2153
- BEY2153 dose 2 (Experimental): Participants administer 26 weeks
  Interventions: Drug: BEY2153
- Placebo (Placebo Comparator): Participants administer 26 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BEY2153 — Participants administer once daily, PO, 26 weeks
  Arms: BEY2153 dose 1; BEY2153 dose 2
Drug: Placebo — Participants administer once daily, PO, 26 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of BEY2153 in patients with early Alzheimer's Disease. Subjects who meet the inclusion and exclusion criteria will be randomized 1:1:1 to one of three treatment arms for 26 weeks administration. The extension study for additional 26 weeks will be conducted open-label with one treatment arm. Subjects will take BEY2153 orally once a day during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults at the age of ≥ 55 to ≤ 85 at the time of informed consent
* Patients diagnosed according to the NIA-AA 2024 Criteria for Diagnosis with Mild Cognitive Impairment (MCI) or diagnosed with mild Alzheimer's disease
* CDR-GS 0.5-1.0 at Screening
* MMSE ≥ 20 at Screening
* Amyloid-positive at amyloid PET scan
* Patients who are capable of understanding information provided and can voluntarily sign written informed consent form

Exclusion Criteria:

* Subjects diagnosed with cognitive impairment due to causes other than substrate causes such as brain lesions, psychiatric disorders, or Alzheimer's disease (e.g., stroke, Parkinson's disease, Lewy body disease, vascular dementia)
* Subjects with any of the following cardiovascular diseases at Screening

  * Cerebrovascular disease within the past 6 months (cerebral infarction, cerebral hemorrhage, transient ischemic attack, etc.)
  * Myocardial infarction or unstable angina pectoris within the past 6 months
  * New York Heart Association (NYHA) Class II congestive heart failure
  * QTcF ≥450 msec or clinically significant electrocardiogram (ECG) abnormalities
* Patients with malignant tumors
* Patients with medical conditions that can affect cognitive decline such as hypothyroidism, vitamin B12 or folate deficiency, niacin deficiency, etc.
* Patients with a history of alcohol related disorders within the past 6 months
* Patients with a positive HIV antibody test result at Screening
* Patients with a positive HBs antigen or HCV antibody test at Screening
* Patients with active bacterial infections who have received antibiotics within 7 days prior to Screening.
* Patients with a history of hypersensitivities to any of the components of investigational product
* Patients who have been hospitalized or treated for suicidal behavior within 5 years prior to Screening or whose C-SSRS results at Screening indicate serious suicidal ideation or behavior
* Patients who have received treatment for Alzheimer's disease (e.g., Lecanemab) within 6 months prior to Screening
* Patients expected to require the administration of a long-acting benzodiazepine (BDZ) for the treatment of sleep disorders at Screening
* Any of the following laboratory test values at Screening:

  * Serum Creatinine >1.5×ULN or eGFR (MDRD) <40 mL/min/1.73 m2
  * Any of the following: AST, ALT >3×ULN, or Total bilirubin >2xULN
* Women who test positive for pregnancy at Screening, or women and men of childbearing potential who are planning to become pregnant, or who do not agree to use adequate contraception* during the study and for 4 weeks after the end of study drug administration

  *Adequate contraception: complete abstinence, hormonal contraceptives with no known drug interactions [Levonorgestrel intrauterine system (IUS) (Mirena), Medroxyprogesterone], surgical sterilization (including vasectomy, bilateral salpingectomy and ligation). However, intermittent abstinence (e.g., using ovulation timing, symptothermal method, or post-ovulation) or external ejaculation are not considered adequate contraception.
* Pregnant or lactating women or women who are tested positive for pregnancy at Screening
* Patients treated with other IP within 4 weeks prior to screening
* Patients who are considered ineligible for study participation for other reasons based on the judgment of the investigator

[Extension Study]

Inclusion Criteria:

* Patients who completed the 26-week visit in the Main Study
* Patients who provided written consent to participate in the Extension Study

Exclusion Criteria:

* Subjects who have dropped out of the Main Study
* Patients who, in the investigator's judgement, are not suitable for participation in Extension Study
* Any of the following laboratory test values at Baseline:

  * Serum Creatinine >1.5×ULN or eGFR (MDRD) <40 mL/min/1.73 m2
  * Any of the following: AST, ALT >3×ULN, or Total bilirubin >2xULN

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Safety: Number of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From Baseline until 4 weeks after the end of treatment

SECONDARY OUTCOMES:
Change from Baseline in Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) after 26-week treatment | Baseline and Week 26
Change from Baseline in Mini Mental State Exam (MMSE) after 26-week treatment | Baseline and Week 26
Change from Baseline in Alzheimer's Disease Assessment Scale-Cognitive 13 (ADAS-Cog 13) after 26-week treatment | Baseline and Week 26
Change from Baseline in Clinician's Interview Based Impression of Change-Plus Caregiver Input (CIBIC-Plus) after 26-week treatment | Baseline and Week 26
Change from Baseline in Alzheimer's Disease Composite Score (ADCOMS) after 26-week treatment | Baseline and Week 26

OTHER OUTCOMES:
Pharmacodynamics: Change in concentrations of plasma AD-related biomarkers | Baseline, Week 6 and Week 26
  To assess the effect of BEY2153 on amyloid (Aβ40, Aβ42) and tau (p-tau217, p-tau181, t-tau) related biomarkers in AD patients
Brain imaging: Change in brain accumulation of amyloid protein | Baseline and Week 26
  Amyloid PET will be conducted following administration of BEY2153 to evaluate the change in brain accumulation of amyloid protein (centiloid)
Brain imaging: Change in brain atrophy | Baseline and Week 26
  vMRI will be conducted following administration of BEY2153 to evaluate the change in brain atrophy (volume)

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Severance Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Yeouido St. Mary's Hospital, Seoul